CLINICAL TRIAL: NCT03509493
Title: Detection of the Common Arrhythmia Atrial Fibrillation in Different Patient Target Groups Using the FibriCheck Smartphone Application
Brief Title: Detection of Atrial Fibrillation in Different Patient Target Groups Using the FibriCheck Smartphone Application
Status: Completed | Type: Observational
Sponsor: Qompium NV (Industry)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2018-04-24; First posted 2018-04-26 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Atrial Fibrillation
Keywords: Primary prevention; Secondary prevention; Clinical practice
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Patients without structural heart disease
  Interventions: Diagnostic Test: FibriCheck
- Patients with structural heart disease
  Interventions: Diagnostic Test: FibriCheck
- Patients with high risk parameters for AF development
  Interventions: Diagnostic Test: FibriCheck
- Patients post-cryptogenic stroke
  Interventions: Diagnostic Test: FibriCheck
- Patients post-cardioversion therapy
  Interventions: Diagnostic Test: FibriCheck
- Patients post-ablation therapy
  Interventions: Diagnostic Test: FibriCheck

INTERVENTIONS:
Diagnostic Test: FibriCheck — Digital health application

SUMMARY:
FibriCheck is a Conformité Européenne (CE)-approved (class IIa) medically diagnostic application that allows for heart rhythm registrations based on an optical signal captured via the smartphone camera. FibriCheck is only available on prescription causing the physician to stay in the 'driving seat' and the application distribution to be traced.

By using FibriCheck, a medically validated smartphone application, daily rhythm measurements can be performed using only the smartphone of the patient. This allows for the heart rhythm to be registered and monitored in a home environment and the data to be automatically sent to the physician. This enables the implementation of FibriCheck in two types of scenarios:

* Scenario 1: the follow-up of patients with high risk parameters for AF development for primary and secondary prevention, whereby detection of AF will result in therapeutic intervention
* Scenario 2: the realisation of monitoring of the heart rhythm of patients post intervention in a home environment

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common heart rhythm disorder affecting 50 million people in Europe and the U.S. It is associated with an increasing mortality and risk for transient cerebrovascular incidents and dementia. De novo AF is in most cases asymptomatic and paroxysmal, causing the diagnosis to be made either by chance or in response to an incident. This drastically impacts the quality of life of the patient and is accompanied with a high socio-economic cost. Guidelines indicate that anticoagulation in patients diagnosed with AF is a cost-effective solution for the prevention of strokes.

In addition, depending on the target group, patients identified with AF can receive therapy in order to control the heart rhythm. These procedures (cardioversion and ablation) often result in follow-up consultations that can be avoided if the heart rhythm can be monitored remotely.

By using FibriCheck, a medically validated smartphone application, daily rhythm measurements can be performed using only the smartphone of the patient. This allows for the heart rhythm to be registered and monitored in a home environment and the data to be automatically sent to the physician. This enables the implementation of FibriCheck in two types of scenarios:

* Scenario 1: the follow-up of patients with high risk parameters for AF development for primary and secondary prevention, whereby detection of AF will result in therapeutic intervention
* Scenario 2: the realisation of monitoring of the heart rhythm of patients post intervention in a home environment

The follow-up of patients is still driven by the treating physician(s). The objective is to implement a correct and successful process management allowing a smooth implementation of "an application on prescription".

Short- and long-term benefits the project wants to prove:

Short-term:

- AF can successfully be detected in a home environment using the FibriCheck application

Long-term: a successful detection of AF in a home environment can:

* Be the first step towards changing and improving the care pathway of the patient
* Induce therapeutic interventions in order to prevent strokes or other complications

ELIGIBILITY:
Inclusion Criteria:

Group 1: Patients without structural heart disease

* Age 65 and older
* CHADSVASc score of 2 or more (including congestive heart failure, hypertension, age, diabetes, previous stroke, vascular disease and sex)
* Comorbidities such as: coronary artery disease, kidney insufficiency, sleep apnea or symptomatic complaints with negative Holter in the past

Group 2: Patients with structural heart disease

* Age 65 and older
* CHADSVASc score of 2 or more
* Left atrial volume indexed for body surface area (BSA) of 34 ml/m² or more, or left atrial diameter > 5 cm
* And any of the following indicators:

  * Diastolic dysfunction of at least grade 2 with restrictive filling (E/A 2 or more) or disturbed relaxation (E/A 0.8) and with E/e' septal 15 or more (E/e' lateral 10 or more) or tricuspid insufficiency (TI) of 2.8 m/s or more
  * At least mitral insufficiency (grade 2/3 or 3/3) or mitral stenosis
  * Hypertrophic (obstructive) cardiomyopathy

Group 3: Patients with high risk parameters for AF development

* Age 65 or more
* General Medical Record in the participating practice
* A 5-year risk of AF of at least 10% according to the CHARGE-AF risk score

Group 4: Patients post-cryptogenic stroke or TIA

- Experienced a cryptogenic TIA or stroke in the past year since the start of the study

Group 5: Patients post-cardioversion therapy

* Confirmed AF patient based on 12-lead ECG
* Successful AF treatment using cardioversion (DCC or chemical) to convert the heart rhythm back to normal sinus rhythm
* Subjects are older than 18 years

Group 6: Patients post-ablation therapy

* Confirmed AF patient based on 12-lead ECG
* Successful AF treatment using ablation therapy to restore the heart rhythm back to sinus rhythm in the past 3 months
* Subjects are older than 18 years

Exclusion Criteria:

* Non-native Dutch
* Pacemaker dependent heart rhythm
* Perniosis patient
* Intense callus formation
* Low adherence to protocol
* Tremor or Parkinson
* Signs of Alzheimer or dementia
* No self-care ability
* Known AF patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients are included in the corresponding group
Sampling Method: Non-Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Detection of unknown atrial fibrillation | 31 December 2017

SECONDARY OUTCOMES:
Detection of recurrent atrial fibrillation | 31 December 2017

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (8):
  - Ziekenhuis Oost Limburg, Genk, Limburg
  - Jessa Ziekenhuis, Hasselt, Limburg
  - AZ Maria Middelares, Ghent, Oost-Vlaanderen
  - AC Huisartsengeneeskunde KU Leuven, Leuven, Vlaams-Brabant
  - HAK Hooglede, Hooglede, West-Vlaanderen
  - Jan Yperman Ziekenhuis, Ieper, West-Vlaanderen
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - AZ Delta Ziekenhuis, Roeselare, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beerten SG, Proesmans T, Vaes B. A Heart Rate Monitoring App (FibriCheck) for Atrial Fibrillation in General Practice: Pilot Usability Study. JMIR Form Res. 2021 Apr 7;5(4):e24461. doi: 10.2196/24461. PMID 33825692